CLINICAL TRIAL: NCT00079157
Title: Phase I Study Of Telomerase Peptide Vaccination For Patients With Advanced Breast Cancer
Brief Title: Vaccine Plus Montanide ISA-51 and Sargramostim in Treating Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000354502; UPCC-11102
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — incomplete Freund's adjuvant; sargramostim

INTERVENTIONS:
Biological: incomplete Freund's adjuvant
Biological: sargramostim
Biological: telomerase: 540-548 peptide vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Giving a vaccine with Montanide ISA-51 and sargramostim may cause a stronger immune response and kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy when given together with Montanide ISA-51 and sargramostim in treating patients with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of telomerase: 540-548 peptide vaccine emulsified in Montanide ISA-51 and sargramostim (GM-CSF) in patients with HLA-A2-expressing stage IV breast cancer.

Secondary

* Compare the generation of human telomerase reverse transcriptase (hTERT) peptide-specific vs cytomegalovirus peptide-specific cytotoxic T-lymphocyte (CTL) immunity in patients treated with this regimen.
* Correlate the dose level of this regimen with the generation of hTERT-specific CTL immunity and the development of hTERT-specific autoimmunity in these patients.
* Determine the tumor response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of the telomerase: 540-548 peptide and CMV 495 peptide portions of the vaccine.

Patients receive telomerase: 540-548 peptide and CMV 495 peptide (as an immunological control) vaccine emulsified in Montanide ISA-51 subcutaneously (SC) followed by sargramostim (GM-CSF) SC on day 1 of weeks 1, 3, 5, 7, 11, 15, 19, and 27 (for a total of 8 vaccinations). Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 5-8 patients receive escalating doses of telomerase: 540-548 peptide and CMV 495 peptide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 5 or 2 of 8 patients experience dose-limiting toxicity. A total of 12 patients receive treatment at the MTD.

Patients are followed within 30 days and then at 6 and 12 months.

PROJECTED ACCRUAL: A total of 5-28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage IV breast cancer
* Failed at least 1 prior conventional therapy for metastatic disease
* Measurable or evaluable disease by clinical, radiographic, or laboratory assessment

  * Measurable lesions must be at least 1 dimension

    * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are not considered measurable:

    * Pleural effusion
    * Bone lesions
    * Tumor markers
* HLA-A2-expressing disease by human leukocyte antigen typing
* No CNS metastases by contrast CT scan and/or MRI

  * No brain metastases within the past 4 years
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* More than 6 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* Hepatitis B negative
* Hepatitis C negative

Renal

* Creatinine ≤ 1.5 times ULN

Immunologic

* HIV negative
* Human T-cell lymphotrophic virus-1 negative
* No active infection
* No major autoimmune disorder that would preclude study participation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No alcohol abuse or illicit drug use within the past 12 months
* No clinically significant comorbid disease or other underlying condition that would preclude study participation
* No significant psychiatric disorder that would preclude giving informed consent or complying with study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior allogeneic or autologous bone marrow or stem cell transplantation
* More than 30 days since prior hematopoietic growth factors
* More than 30 days since initiation of prior immunotherapy (e.g., trastuzumab [Herceptin])
* Concurrent immunotherapy (e.g., trastuzumab) allowed provided regimen was initiated more than 30 days before study entry, disease is stable or progressive, and patient plans to continue immunotherapy for the duration of study participation
* No other concurrent hematopoietic growth factors

Chemotherapy

* More than 30 days since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* More than 30 days since prior glucocorticoids
* More than 30 days since initiation of prior hormonal therapy (e.g., tamoxifen, anastrozole, or letrozole)
* Concurrent hormonal therapy (e.g., tamoxifen, anastrozole, or letrozole) allowed provided regimen was initiated more than 30 days before study entry, disease is stable or progressive, and patient plans to continue hormonal therapy for the duration of study participation
* No concurrent glucocorticoids

Radiotherapy

* More than 30 days since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 14 days since prior anticoagulants (e.g., warfarin, heparin, or enoxaparin)

  * Low-dose anticoagulants to maintain IV catheter patency allowed
* More than 30 days since prior immunosuppressive drugs
* More than 30 days since prior experimental therapy
* No concurrent immunosuppressive drugs
* No other concurrent investigational products

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2004-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Domchek, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States